CLINICAL TRIAL: NCT06106126
Title: Pharmacokinetics and Safety of GST-HG171 Tablets in Subjects With Impaired and Normal Renal Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Akeylink Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GST-HG171-I-03
Record Dates: First submitted 2022-12-29; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2022-12

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mild renal impairment (Other)
  Interventions: Drug: GST-HG171 Tablets
- Moderate renal impairment (Other)
  Interventions: Drug: GST-HG171 Tablets
- Severe renal impairment (Other)
  Interventions: Drug: GST-HG171 Tablets
- Normal Renal Function (Other)
  Interventions: Drug: GST-HG171 Tablets

INTERVENTIONS:
Drug: GST-HG171 Tablets — 150mg GST-HG171 100mg Tablets and ritonavir

SUMMARY:
This si a single-center, non-randomized, open, parallel, single-dose trial was designed to evaluate the safety and pharmacokinetic characteristics of GST-HG171 tablets in subjects with impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to meet all of the following conditions

1. Voluntarily sign informed consent prior to the start of activities related to this study, be able to understand the procedures and methods of this study, and be willing to strictly follow the clinical trial protocol to complete this study;
2. Subjects (including their partners) are willing to have no family planning and voluntarily take highly effective contraception within 6 months after the last study drug administration;
3. Age range from 18 to 70 (including both ends) on the date of signing the informed consent, both male and female;
4. Male subjects weigh at least 50 kg and female subjects weigh at least 45 kg; Body mass index (BMI) 18-32 kg/m2 (including both ends);

   Subjects with normal renal function should also meet all of the following conditions:
5. Physical examination, vital signs and electrocardiogram are normal or abnormal without clinical significance;
6. The glomerular filtration rate should meet the following criteria: Subjects with normal renal function: GFR≥90 mL/min;
7. The following demographic matching criteria must be met during screening:

   1. The body weight was matched with that of the renal impairment group, with an average of ±10 kg;
   2. Age matching was performed with the renal impairment group, with the mean ±10 years old;
   3. Gender matching was performed with the group of renal impairment, with the mean ±1 case;

   Subjects with renal impairment should also meet all of the following conditions:
8. Have chronic kidney disease (CKD), have any indicators of kidney injury or have a GFR less than 60 mL/min for more than 3 months (outpatient medical records, inpatient records or laboratory records can be used as evidence);
9. The glomerular filtration rate shall meet the following criteria: Subjects with mild renal impairment (stage CKD2) : 60-89 mL/min (including values at both ends), subjects with moderate renal impairment (stage CKD3) : 30-59 mL/min (including values at both ends), subjects with severe renal impairment (stage CKD4) : 15-29 mL/min (including both ends);
10. Renal function was stable, and GFR results of two tests before administration (at least 3 days apart) should be in the same CKD stage;
11. Except for renal dysfunction and complications, the investigator judged that the physical condition was good based on medical history inquiry, comprehensive physical examination, routine laboratory examination (blood routine, blood biochemistry, urine routine, coagulation function, etc.), 12-lead electrocardiogram, chest X-ray (orthographic), abdominal B-ultrasound examination, etc.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will not be enrolled in this study

1. Allergic constitution, including severe drug allergy or history of drug allergy, known allergy to the study drug or any component of the study drug;
2. Those who donated blood ≥400 mL within 3 months before screening, or donated blood ≥200 mL within 1 month before screening, or received blood transfusion or used blood products;
3. Patients with severe infection, trauma, gastrointestinal surgery or other major surgical operations within 4 weeks before screening;
4. A history of difficulty swallowing or any gastrointestinal disorder affecting drug absorption, including frequent nausea or vomiting due to any etiology;
5. A strong or medium acting inducer or inhibitor of CYP3A enzyme, a strong P-gp inhibitor or P-gp inducer used within 1 month before screening;
6. Those who had been vaccinated within 14 days prior to screening or planned to be vaccinated during the study period;
7. Smokers who smoked at least 10 cigarettes a day in the 3 months before screening;
8. had taken a special diet (including dragon fruit, mango, grapefruit, and/or xanthine diet, chocolate) and/or had consumed excessive amounts of tea, coffee, grapefruit/grapefruit juice and/or caffeinated beverages (more than 8 cups of 200 mL per cup per day on average) in the 2 weeks prior to administration;
9. A history of drug or substance abuse and/or alcoholism (14 units of alcohol per week: 1 unit = 285 mL for beer, 25 mL for spirits, or 100 mL for wine);
10. had taken any products containing alcohol or had tested positive for alcohol breath test within 24 hours before receiving the study drug;
11. Positive urine drug screening (morphine, cannabis);
12. Pregnant or lactating women or women of childbearing age who have tested positive for pregnancy;
13. Active HBV or HCV infection, HIV-positive, or treponema pallidum antibody positive and rapid plasma response (RPR) positive (RPR only for treponema pallidum antibody positive);
14. Those not suitable for inclusion for other reasons;

    Subjects with normal renal function should be excluded if they meet any of the following exclusion criteria:
15. Participants who have participated in clinical trials of drugs or medical devices within 3 months prior to screening (subject to drug acceptance);
16. had taken any prescription drugs, over-the-counter drugs, any vitamin products or herbs in the 14 days prior to screening;
17. Abnormal clinical laboratory examination with clinical significance, or other clinically significant diseases (including but not limited to respiratory system, digestive system, urinary system, nervous system, blood system, endocrine system, tumor, immune, psychiatric or cardiovascular and cerebrovascular diseases) found by other clinical findings in the 12 months prior to screening;

    Subjects with renal impairment should be excluded if they meet any of the following exclusion criteria:
18. Participants who have participated in clinical trials of drugs or medical devices within 1 month before screening (subject to drug acceptance);
19. Patients with acute renal failure or who have had a kidney transplant; Or require kidney dialysis during the study;
20. In addition to the chronic primary renal disease itself and its complications, those who have suffered from or currently suffer from other serious systemic organ diseases, including but not limited to digestive system, respiratory system, nervous system, blood system, endocrine system, tumor, immune system, psychiatric or cardiovascular and cerebrovascular diseases, and are judged by the study doctor as unfit to participate in this study;
21. hypertension that is not well controlled by antihypertensive medications (systolic blood pressure ≥150 mm Hg or diastolic blood pressure ≥100 mm Hg);
22. Laboratory examination: alanine aminotransferase (ALT) ≥2×ULN, aspartate aminotransferase (AST) ≥2×ULN; Serum total bilirubin >1.5×ULN; Albumin <30 g/L; Neutrophil absolute value <1.3×109/L; Hemoglobin <60g/L; Platelet count <100×109/L;
23. New York Heart Association (NYHA) Grade III or IV for congestive heart failure, or left ventricular ejection fraction <50% at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for GST-HG171 | Day 1 (predose), 0.25,0.5 ,0.75,1 ,1.25,1.5,2 ,3 ,4 ,6 ,8 ,12,24 ,48 and 72 hours post-dose
  Maximum observed plasma GST-HG171 concentration.

SECONDARY OUTCOMES:
AEs | up to Day 10
  To evaluate the safety and tolerability of GST-HG171 tablets in subjects with impaired renal function.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided